CLINICAL TRIAL: NCT03469765
Title: (TIMP-2)x(IGFPB7) as Early Renal Biomarker for the Prediction of Acute Kidney Injury in Aortic Surgery - an Observational Study (TIGER)
Brief Title: (TIMP-2)x(IGFPB7) to Predict Acute Kidney Injury (AKI) in Aortic Surgery
Acronym: TIGER
Status: Completed | Type: Observational
Sponsor: Jörg Schefold (Other)
Responsible Party: Sponsor-Investigator, Jörg Schefold, Sponsor-investigator, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: TIGER
Record Dates: First submitted 2018-03-09; First posted 2018-03-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Renal Failure; Dialysis; Aortic Surgery; Biomarker; Acute Kidney Injury
Keywords: AKI
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of patients after aortic surgery: with subanalysis of patients with/without supra-/infrarenal surgery
  Interventions: Other: does not apply

INTERVENTIONS:
Other: does not apply — biological sample taking: urine, blood

SUMMARY:
New biomarkers that predict the development of renal dysfunction in patients with aortic surgery are urgently needed. The investigators investigate whether urinary (TIMP-2)x(IGFBP7) predicts postoperative Acute Kidney Injury and/or need for Renal Replacement Therapy (RRT) in patients after aortic surgery (including EVAR).

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of emergency or elective abdominal aortic surgery (infra- or suprarenal clamping or EVAR) are eligible for study inclusion.

Exclusion Criteria:

* Patients unable to give informed consent
* Age < 18
* Patients not speaking German or French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with need for aortic operation/ repair
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Statistically significant difference in mean total (TIMP-2)x(IGFBP7) values of patients with/ without AKI (as defined along Kidney Disease Initiative for Improvement of global outcomes (KDIGO) definitions: stages 1-3) at the first postoperative day. | 24 hours following ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Waskowski J, Pfortmueller CA, Schenk N, Buehlmann R, Schmidli J, Erdoes G, Schefold JC. (TIMP2) x (IGFBP7) as early renal biomarker for the prediction of acute kidney injury in aortic surgery (TIGER). A single center observational study. PLoS One. 2021 Jan 7;16(1):e0244658. doi: 10.1371/journal.pone.0244658. eCollection 2021. PMID 33411755